CLINICAL TRIAL: NCT07301242
Title: Population Pharmacokinetic/Pharmacodynamic Modeling of Ciprofol in Elderly Patients Undergoing Orthopedic Limb Surgery
Brief Title: Population Pharmacokinetics and Pharmacodynamics of Ciprofol
Status: Recruiting | Type: Observational
Sponsor: Shanghai Geriatric Medical Center (Other)
Responsible Party: Principal Investigator, Xue Zhang, Attending Physician, Shanghai Geriatric Medical Center
Other Study IDs: ZCLY2025-021
Record Dates: First submitted 2025-11-19; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-11

CONDITIONS: Hip Fractures (ICD-10 72.01-72.2); Osteoarthritis, Knee and Hip; Femoral Neck Fractures
MeSH Terms: conditions — Hip Fractures; Osteoarthritis; Femoral Neck Fractures | interventions — (2-(1R)-1-cyclopropyl)ethyl-6-isopropyl-phenol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood and plasma samples will be retained for pharmacokinetic and pharmacodynamic analysis. No DNA extraction will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Elderly Orthopedic Limb Surgery Cohort: Inclusion Criteria:
  Age ≥65 years; BMI 18-30 kg/m²; ASA physical status classification I-III; Scheduled for elective orthopedic limb surgery under general anesthesia; Expected duration of surgery >30 minutes; Willing to participate and able to provide written informed consent.
  Exclusion Criteria:
  Known allergy to ciprofol or related medications, or any contraindication to their use; Preoperative cognitive impairment (Mini-Cog score <3); History of severe cerebrovascular disease or related complications; History of neuromuscular system diseases or psychiatric disorders; History of sedative medication use; History of alcohol abuse or substance use disorder; Bradycardia (heart rate <60 beats per minute); Hypotension (mean arterial pressure <55 mmHg); QT interval prolongation; Uncooperative or unable to communicate effectively.
  Interventions: Drug: Ciprofol

INTERVENTIONS:
Drug: Ciprofol — Ciprofol is used as an intravenous anesthetic agent for sedation and anesthesia induction/maintenance in elderly patients undergoing elective orthopedic limb surgery. In this observational study, ciprofol is administered according to standard clinical practices, and data on its pharmacokinetics, pharmacodynamics, safety, and effectiveness in this specific population will be collected.
  Other Names: Cipepofol; Sishuning

SUMMARY:
The goal of this observational study is to learn how the anesthetic drug ciprofol works in older adults who are having limb surgery under general anesthesia at Shanghai Geriatric Medical Center. The study will help researchers build a population model to better understand how the drug moves through the body (PK) and how it affects patients (PD). This model may help doctors use a Target-Controlled Infusion (TCI) system to adjust the drug dose more precisely.

The main question it aims to answer is: Does ciprofol work safely and effectively in older adults during orthopedic surgery?

Participants already receiving ciprofol as part of their regular anesthesia care will:

1. Provide blood samples at different time points during and after surgery.
2. Have their vital signs and anesthesia-related data recorded before, during, and after surgery.
3. Be monitored for side effects and recovery indicators such as the Aldrete score and signs of postoperative delirium.

Researchers will use this information to:

1. Build and test a population PK/PD model for ciprofol.
2. Simulate recommended TCI dosing plans.
3. Explore how individual responses to ciprofol relate to recovery and safety outcomes.

This study may help improve anesthesia care for elder adults by making drug dosing safer and more effective.

DETAILED DESCRIPTION:
Elderly patients undergoing orthopedic limb surgery represent a growing population with unique perioperative challenges. Age-related physiological changes-including reduced hepatic and renal function, altered body composition, and decreased cardiac output-significantly affect the pharmacokinetics (PK) and pharmacodynamics (PD) of anesthetic drugs. These changes increase the difficulty of maintaining adequate anesthesia depth and hemodynamic stability.

Ciprofol, a novel intravenous anesthetic, has shown promising efficacy and safety in clinical practice. However, existing PK/PD models are largely derived from healthy volunteers or younger patients, and cannot adequately predict drug behavior in elderly orthopedic patients who often present with comorbidities and heightened surgical stress. This gap may lead to risks such as drug accumulation and circulatory depression, or insufficient dosing and intraoperative awareness.

This single-center, observational, prospective study at Shanghai Geriatric Medical Center aims to construct and validate a population PK/PD model of ciprofol specifically for elderly patients undergoing orthopedic limb surgery. The model will support precise control of effect-site concentration via Target-Controlled Infusion (TCI) systems, enabling individualized anesthesia management.

Study Objectives 1.Primary Objective: To develop and validate a population PK/PD model of ciprofol tailored to elderly orthopedic patients, and to evaluate its accuracy in predicting effect-site concentrations.

2.Secondary Objectives:

1. To simulate recommended TCI dosing regimens based on the new model and compare them with current drug label recommendations, assessing clinical value and optimization potential.
2. To evaluate the anesthetic efficacy and safety of ciprofol in this patient population.

3.Exploratory Objectives: To investigate the influence of covariates (e.g., age, sex, BMI, hepatic and renal function) on PK/PD parameters, and to explore correlations between individual PK/PD parameters and recovery outcomes such as Aldrete score and postoperative delirium incidence.

Study Design

1.Type: Single-center, observational, biosample-utilization study. 2.Population: 45 elderly patients (≥65 years, ASA I-III) scheduled for elective orthopedic limb surgery under general anesthesia.

3.Procedures:

1. Collection of perioperative clinical data (vital signs, BIS monitoring, anesthesia-related indicators).
2. Serial blood sampling at predefined time points for plasma concentration measurement.
3. Monitoring of anesthetic efficacy (induction success, BIS values, recovery times) and safety endpoints (hypotension, bradycardia, hypoxemia, injection pain).

4.Endpoints:

1. Primary Endpoint: Accuracy of the population PK/PD model in predicting effect-site concentrations.
2. Secondary Endpoints: Differences between model-recommended dosing and label-based dosing; incidence of ciprofol-related adverse events; anesthetic efficacy indicators.
3. Exploratory Endpoints: Covariate effects on PK/PD parameters; correlation of PK/PD parameters with Aldrete score recovery and postoperative delirium.

Data Management and Analysis All perioperative data will be recorded and stored electronically, with double-entry verification and query resolution procedures to ensure accuracy. PK/PD modeling will be performed using nonlinear mixed-effects modeling (NONMEM). Model evaluation will include goodness-of-fit plots, visual predictive checks, and bootstrap validation. Simulations will be conducted to compare TCI dosing regimens derived from the new model with standard recommendations.

Expected Significance This study will fill an important gap in anesthetic pharmacology by providing a validated PK/PD model of ciprofol for elderly orthopedic patients. The findings are expected to improve perioperative anesthesia management, enhance patient safety, and support individualized dosing strategies in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years;
* BMI: 18-30 kg/m²;
* ASA physical status classification I-III;
* Scheduled for elective orthopedic limb surgery under general anesthesia;
* Expected duration of surgery >30 minutes;
* Willing to participate and able to provide written informed consent.

Exclusion Criteria:

* Known allergy to ciprofol or related medications, or any contraindication to their use;
* Preoperative cognitive impairment;
* History of severe cerebrovascular disease or related complications;
* History of neuromuscular system diseases or psychiatric disorders;
* History of sedative medication use;
* History of alcohol abuse or substance use disorder;
* Bradycardia (heart rate <60 beats per minute);
* Hypotension (mean arterial pressure <55 mmHg);
* QT interval prolongation;
* Uncooperative or unable to communicate effectively.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients undergoing orthopedic limb surgery
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-10-28 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Plasma Concentration of Ciprofol | From the start of drug administration to 24 hours after the end of drug administration.
  Arterial or venous blood samples (1 mL each) will be collected to measure the plasma concentration of ciprofol using liquid chromatography - mass spectrometry. These concentration data points will be used to construct the population pharmacokinetic model. Reported in ng/mL.
Bispectral Index (BIS) Value | Continuously monitored from the start of anesthesia induction, throughout the maintenance phase, until full recovery (approximately up to 4 hours).
  The BIS value is a non-invasive measure of the level of consciousness/depth of anesthesia, ranging from 0 (isoelectric EEG) to 100 (awake). It is used as the pharmacodynamic metric for modeling.
Modified Observer's Assessment of Alertness/Sedation (MOAA/S) Score | Induction phase (every minute until loss of consciousness); Maintenance phase; and Post-operative phase (every 3 minutes in PACU until score returns to 5), up to approximately 4 hours.
  The MOAA/S scale is a categorical measure used to assess the depth of sedation/anesthesia. Scores range from 0 (No response to painful stimulus) to 5 (Responds readily to name spoken in normal tone). This metric will be used as a pharmacodynamic endpoint to construct a categorical PK/PD model (e.g., proportional odds model) relating ciprofol concentration to clinical sedation depth.

SECONDARY OUTCOMES:
Mean Arterial Pressure (MAP) | Continuously measured during the induction, maintenance (intra-operative), and recovery phase (up to 2 hours post-infusion).
  Evaluation of hemodynamic stability by measuring the absolute value of Mean Arterial Pressure. Reported in millimeters of mercury (mmHg).
Heart Rate | Continuously measured during the induction, maintenance (intra-operative), and recovery phase (up to 2 hours post-infusion).
  Evaluation of hemodynamic stability by measuring the absolute value of Heart Rate. Reported in beats per minute (bpm).

CONTACTS AND LOCATIONS:
Overall Officials: Xue Zhang, Principal Investigator — Shanghai Geriatric Medical Center
Locations (1):
- Shanghai Geriatric Medical Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No